CLINICAL TRIAL: NCT06745518
Title: A Phase 2, Randomized, Placebo-controlled, Double-blind, Phosphate Binder-combination Study of TS-172 in Hyperphosphatemia Patients on Hemodialysis
Brief Title: A Phase 2 Study of TS-172 in Hyperphosphatemia Patients on Hemodialysis With Phosphate Binders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TS172-02-03
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Hyperphosphatemia Patients on Hemodialysis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TS-172 (Experimental)
  Interventions: Drug: TS-172
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TS-172 — oral administration of TS-172 20~60 mg/day
  Arms: TS-172
Drug: Placebo — oral administration of placebo
  Arms: Placebo

SUMMARY:
A phase 2, randomized, placebo-controlled, double-blind, phosphate binder-combination study of TS-172 in hyperphosphatemia patients on hemodialysis

ELIGIBILITY:
Inclusion Criteria:

1. Hyperphosphatemia patients (outpatients) with chronic kidney disease receiving hemodialysis (HD or HDF) 3 times a week for at least 12 weeks prior to Visit 1 (Week -3)
2. Patients aged >= 18 years at the time of obtaining informed consent
3. Patients with a serum phosphorus concentration of >= 5.5 mg/dL and < 10.0 mg/dL at Visit 1 (Week -3)
4. Patients who have been prescribed at least one phosphate binder within the approved dosage, and the prescribed drug and dosage regimen should have been unchanged during the last 2 weeks prior to Visit 1 (Week -3)

Exclusion Criteria:

1. Patients with confirmed serum intact PTH concentration >500 pg/mL from Visit 1 (Week -3) to Visit 4 (Week 0)
2. Patients who have undergone previous parathyroid intervention (PTx, PEIT, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Achievement rate of the target serum phosphorus level | Week 8

SECONDARY OUTCOMES:
Change from baseline in serum concentration of phosphorus | Up to Week 8
Concentration of corrected serum calcium | Up to Week 8
Serum Ca × P product | Up to Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Taisho Director, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No